CLINICAL TRIAL: NCT07401134
Title: Improving Postoperative Recovery: A Randomized Study of Multimodal Perineal Analgesia Protocol (MPAP) After Vaginal Surgery
Brief Title: Improving Postoperative Recovery: A Study of Multimodal Perineal Analgesia Protocol (MPAP) After Vaginal Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Katherine Amin, Assistant Professor of Clinical Urology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20251232
Record Dates: First submitted 2026-01-28; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Perineal Injury; Pain Vulva; Perineum; Injury
MeSH Terms: conditions — Vulvodynia; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Perineal Analgesic Protocol (MPAP) (Experimental): Participants will follow the Multimodal Perineal Analgesic Protocol (MPAP) in addition to their normal post-operation care. Participants will receive a Perineal Care Kit prior to discharge from the hospital. This kit will contain:
  * 14 perineal ice packs
  * One container of 100 medicated witch-hazel pads (MAJOR® Medi-Pads)
  * One 2.75 oz can of 20% benzocaine with aloe spray (Dermoplast®)
  Participants will also receive standard discharge instructions, including guidance on perineal hygiene, scheduled pain relievers, activity restrictions, constipation prevention, and catheter care if a catheter has been placed.
  Interventions: Drug: Perineal ice packs, medicated witch-hazel pads, and topical benzocaine spray
- Normal Post-Operation Care (No Intervention): Participants will receive standard discharge instructions, including guidance on perineal hygiene, scheduled pain relievers, activity restrictions, constipation prevention, and catheter care if a catheter has been placed.

INTERVENTIONS:
Drug: Perineal ice packs, medicated witch-hazel pads, and topical benzocaine spray — Participants will follow the Multimodal Perineal Analgesic Protocol (MPAP) in addition to their normal post-operation care. Participants will receive a Perineal Care Kit prior to discharge from the hospital. This kit will contain 14 perineal ice packs, one container of 100 medicated witch-hazel pads (MAJOR® Medi-Pads), and one 2.75 oz can of 20% benzocaine with aloe spray (Dermoplast®). Participants will receive written instructions for use of these products.
  Arms: Multimodal Perineal Analgesic Protocol (MPAP)

SUMMARY:
The purpose of this research is to determine if using perineal ice packs, medicated witch-hazel pads (MAJOR® Medi-Pads), and topical benzocaine spray (Dermoplast®) helps reduce perineal pain after perineorrhaphy and/or posterior colporrhaphy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* Undergoing perineorrhaphy and/or posterior colporrhaphy (rectocele repair/posterior repair) as part of their planned vaginal pelvic reconstructive surgery
* Physically able to apply medicated witch-hazel pads (MAJOR® Medi-Pads) and administer topical benzocaine spray (Dermoplast®) to the perineal area
* Able to understand and willing to provide informed consent

Exclusion Criteria:

* Known allergy or hypersensitivity to any of the study products or components, including witch hazel, benzocaine, aloe, or other product ingredients
* Minors
* Presence of an indwelling catheter expected to remain in place for ≥7 days postoperatively
* History of chronic pelvic pain syndromes that may confound postoperative pain assessment, including interstitial cystitis/bladder pain syndrome (IC/BPS), endometriosis, pudendal neuralgia, or vulvodynia
* Chronic use (> 3 weeks of continuous use) of opioid pain medication
* Presence of vulvar dermatoses such as lichen sclerosus, lichen planus, or lichen simplex chronicus
* Currently pregnant or breastfeeding
* Anticipated inability to complete postoperative follow-up, including physical or cognitive limitations that would impede self-care or completion of study diaries
* Inability or unwillingness to provide informed consent or comply with study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Difference in Perineal Pain Score on Postoperative Day (POD) 3 Between Control and Interventional Groups | 3 Days
  Perineal Pain Score will be assessed using a 10-cm Visual Analog Scale (VAS). It consists of a 10 cm line with "no pain" at one end (0) and "worst possible pain" at the other (10). Participants will mark the line to indicate their level of pain or sensation. A higher score indicates a more severe level of pain.

SECONDARY OUTCOMES:
Difference in Daily Pain Scores Within Post-Operative Days 0-7 Between Control and MPAP Groups | 7 Days
  Pain Score will be assessed using a continuous 10-cm Visual Analog Scale (VAS). It consists of a linear scale with "no pain" at one end (0) and "worst possible pain" at the other (10). To use it, the patient marks the line to indicate their level of pain or sensation. A higher score indicates a more severe level of pain. Daily VAS values will be plotted on a pain-time graph, and will be compared using a mixed-effects model for repeated measures.
Difference in Total Number of Doses of Each Class of Analgesic Medications Within Post-Operative Days 0-7 Between Control and Interventional Groups | 7 Days
  The number of doses and class of analgesic medication (acetaminophen, NSAIDs, or opioids) will be recorded in a medication diary for control and interventional groups on post-operative days 0-7. A higher number of doses will be interpreted to higher pain burden.
Difference in Patient Satisfaction Scores at 2 Weeks Post-Operation Between Control and Interventional Groups | 2 Weeks
  Patient satisfaction with pain management will be measured using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied) at the 2-week postoperative visit. Median scores will be calculated for control and interventional groups. A lower value will indicate lower satisfaction while higher scores indicate higher satisfaction.
Incidence of Adverse Events Experienced by Participants Within Post-Operative Days 0-7 Between Control and Interventional Groups | 7 Days
  Proportion of participants in each study group (control and intervention) who experience any local adverse reaction, including rash, burning, itching, or irritation, at the application site. Reactions will be recorded in participant daily diaries and/or reported during follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Amin, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Hospitals and Clinics, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No